CLINICAL TRIAL: NCT05096884
Title: Post-Acute Sequelae of Coronavirus-19 (COVID-19) With DysPnEA on ExertIon And Associated TaChycardia TrEatment Study
Acronym: PEACE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021-1100
Record Dates: First submitted 2021-10-25; First posted 2021-10-27 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Tachycardia; Dyspnea; COVID-19
Keywords: COVID-19; Post-COVID; Long-COVID; Tachycardia; Shortness of breath; Post-Acute Sequelae of COVID-19 (PASC)
MeSH Terms: conditions — Tachycardia; Dyspnea; COVID-19; Post-Acute COVID-19 Syndrome | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm - Metoprolol Succinate. (Experimental): The beta blocker metoprolol succinate will be initiated at a starting low dose of 25 mg daily for two weeks and will be escalated if well tolerated every 2 weeks to a maximum dose of 400 mg po daily.
  Interventions: Drug: Metoprolol Succinate

INTERVENTIONS:
Drug: Metoprolol Succinate — The beta blocker metoprolol succinate will be initiated at a starting low dose of 25 mg daily for two weeks and will be escalated if well tolerated every 2 weeks to a maximum dose of 400 mg po daily.

SUMMARY:
Most patients with acute COVID-19 (Coronavirus 19) recover within weeks, however a significant number of individuals will develop the post-acute COVID 19 syndrome (PASC). As of July 2021, the post COVID syndrome qualifies as a disability under the Americans with Disabilities Act. The symptoms which comprise this condition are highly variable and often extraordinarily debilitating. They may be distinct from the initial presentation or may mimic those which defined the initial infection. The post COVID syndrome can be diagnosed when symptoms persist longer than 3 months and may extend to beyond one year. There are risks for permanent levels of disability. Patients who seemingly did not have active COVID-19 symptoms in the days following infectious exposure may also develop post Covid syndromes. These syndromes are considered to constitute a distinct clinical entity which has of yet no clearly defined pathogenic mechanism or validated treatment algorithms.

International investigative efforts are now underway to determine who might develop the post COVID syndrome, it's long term consequences and how best to treat its many problematic symptoms.

DETAILED DESCRIPTION:
Although the long Covid syndrome or PASC is a well recognized syndrome, its pathogenesis is poorly understood. Hypotheses have included persistent viral remnants with consequent provocation of the generalized symptoms characteristic of systemic inflammation. The virus may continue to infect heart, lung or neurologic tissue rendering various organs dysfunctional. Alternatively there could be persistently infected or damaged endothelial cells which line blood vessels and thereby create perturbations of blood flow.

The altered blood flow might then explain the many reported symptoms. However the pathogenesis can be distinguished and studied independently from the physiological disturbance. Existing and accepted therapies for tachycardia and shortness of breath, although they might not reverse the virus caused injury, could be used to reduce the resultant physiologic abnormalities which in turn produce the symptoms of the long Covid syndrome. Beta blockers are standard therapies in sinus tachycardias, (1,2) and postural orthostatic tachycardia syndrome (POTS) (3,4) which are often characterized by high levels of sympathetic drive which beta blockers are designed to modulate.

Thus it is reasonable to hypothesize that that treatment with beta blockers may be an effective intervention as Covid-19 directly infects the nerve and vascular tissues which regulate sympathetic excess which in turn may produce the cardiovascular symptoms of PASC. Moreover it is important to specifically study beta blockers in PASC because they are currently actively in use for this indication. Yet the possibility remains that although the symptoms are similar to those in which beta blockers have been effective, the pathologic processes in PASC will not be responsive to beta blocker therapy. If this were to be true, beta blockers would prove ineffective and might carry a risk of harm. Equally as important is to properly determine the effective dose as the therapeutic window for these agents is wide.

Metoprolol which is a widely used agent in cardiovascular disease is approved in doses ranging from 25 to 400 mg per day. The proposed study will compare 6 minute walk distances (pre and post the treatment), the echocardiographic measurement of the impact of sympathetic excess on the heart's ability to empty effectively and a quality of life survey. Each of these study elements will be measured before and after progressively increased doses of beta blocker.

Our study is thus designed to study two issues:

1. Whether beta blockers which have been utilized to treat tachycardias, POTS (postural orthostatic tachycardia syndrome), and hypertension will have similar effectiveness in PASC
2. To determine appropriate dosing which may be different than those used on non PASC conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject should be between the ages of 18 and 40 with DOE (dyspnea on exertion) for 3 - 12 months
2. Subjects recovered from acute, polymerase chain reaction (PCR) positive, COVID-19 infection
3. Recovery from COVID-19 will be defined as substantial improvement in or essential resolution of initial clinical symptoms
4. Demonstration of tachycardia and/or dyspnea with minimal activity (subjectively different than pre-COVID 19 infection state)
5. Abnormal HUTT (heads up tilt test)
6. Normal chest x-ray
7. Left ventricular ejection fraction (LVEF) >50% by transthoracic echocardiography
8. Zva >3.5 as calculated from TTE (transthoracic echocardiogram).
9. Hemoglobin/Hematocrit within normal laboratory standards
10. Thyroid-stimulating hormone (TSH) within normal laboratory standards

Exclusion Criteria:

1. Active pregnancy (negative pregnancy test is the standard of care prior to HUTT)
2. Demonstrate a primary cause of appropriate DOE and sinus tachycardia

   1. Fevers/infection
   2. Hypovolemia
   3. Anemia
   4. Hyperthyroidism
   5. Alcohol/drug/medication withdrawal
3. Currently taking beta blocker medications
4. Currently being treated for pre-existing neurally mediated hypotension/syncope or known dysautonomia.
5. Medical history of chronic lung disease or reactive airway syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Landers, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page RL, Joglar JA, Caldwell MA, Calkins H, Conti JB, Deal BJ, Estes NA 3rd, Field ME, Goldberger ZD, Hammill SC, Indik JH, Lindsay BD, Olshansky B, Russo AM, Shen WK, Tracy CM, Al-Khatib SM; Evidence Review Committee Chairdouble dagger. 2015 ACC/AHA/HRS Guideline for the Management of Adult Patients With Supraventricular Tachycardia: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2016 Apr 5;133(14):e506-74. doi: 10.1161/CIR.0000000000000311. Epub 2015 Sep 23. No abstract available. PMID 26399663
- [Background] Brugada J, Katritsis DG, Arbelo E, Arribas F, Bax JJ, Blomstrom-Lundqvist C, Calkins H, Corrado D, Deftereos SG, Diller GP, Gomez-Doblas JJ, Gorenek B, Grace A, Ho SY, Kaski JC, Kuck KH, Lambiase PD, Sacher F, Sarquella-Brugada G, Suwalski P, Zaza A; ESC Scientific Document Group. 2019 ESC Guidelines for the management of patients with supraventricular tachycardiaThe Task Force for the management of patients with supraventricular tachycardia of the European Society of Cardiology (ESC). Eur Heart J. 2020 Feb 1;41(5):655-720. doi: 10.1093/eurheartj/ehz467. No abstract available. PMID 31504425
- [Background] Deng X, Zhang Y, Liao Y, Du J. Efficacy of beta-Blockers on Postural Tachycardia Syndrome in Children and Adolescents: A Systematic Review and Meta-Analysis. Front Pediatr. 2019 Nov 7;7:460. doi: 10.3389/fped.2019.00460. eCollection 2019. PMID 31788462
- [Background] Raj SR, Black BK, Biaggioni I, Paranjape SY, Ramirez M, Dupont WD, Robertson D. Propranolol decreases tachycardia and improves symptoms in the postural tachycardia syndrome: less is more. Circulation. 2009 Sep 1;120(9):725-34. doi: 10.1161/CIRCULATIONAHA.108.846501. Epub 2009 Aug 17. PMID 19687359

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Arm - Metoprolol Succinate.
Started | 14
Completed | 10
Not Completed | 4
Not completed — Excluded based on negative tilt table test | 4

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm - Metoprolol Succinate.
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 42.5 [20 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Walk Test at the End of Treatment Period
Description: To assess the reduction of symptoms in patients with PASC Dyspnea on Exertion (DOE) and associated tachycardia when treated with beta blockers as captured in patients walk test. Walk test will be performed at day 1 (baseline) and at 2-4 weeks post treatment completion which consists of 8 weeks metoprolol succinate (approximately 12 weeks from baseline).
Time Frame: 12 weeks from baseline walk test
Population: Total distance walked within 6 minutes
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Study Arm - Metoprolol Succinate.
Number analyzed (Participants) | 10
meters
  Distance walked at baseline | 275 (76)
  Distance walked post treatment | 339 (76)

2. Primary Outcome: Change in Zva Measurement at the End of Treatment Period
Description: To assess the reduction of symptoms in patients with PASC Dyspnea on Exertion (DOE) and associated tachycardia when treated with beta blockers as captured in Zva measurement calculated from patient's TTE (transthoracic echocardiogram).
  TTE (and Zva) will be performed at day 1 (baseline) and at 2-4 weeks post treatment completion which consists of 8 weeks metoprolol succinate (approximately 12 weeks from baseline).
Time Frame: 12 weeks from baseline transthoracic echocardiogram (TTE).
Population: Zva measurement in (mmHg mL^-1) m^2
Measure: Mean (Standard Deviation); unit: (mmHg mL^-1) m^2
Arm/Group | Study Arm - Metoprolol Succinate.
Number analyzed (Participants) | 10
(mmHg mL^-1) m^2
  Zva at baseline | 4.24 (0.83)
  Zva post treatment | 3.70 (0.72)

3. Secondary Outcome: Change in Minnesota Living With Heart Failure Score at the End of Treatment Period
Description: Subjective improvement in Dyspnea on Exertion (DOE), tachycardia and well being score as measured by the Minnesota Living with Heart Failure.
  The Minnesota Living with Heart Failure questionnaire will be administered at day 1 (baseline) and at 2-4 weeks post treatment completion which consists of 8 weeks metoprolol succinate (approximately 12 weeks from baseline). Minnesota Living with Heart Failure questionnaire is a 21-item questionnaire with each item having a 6 point Likert scale (0-5), Zero represents "No symptom" and 5 represents high intensity of symptom. The questionnaire has 3 dimension and they measure Physical, socio-economic and emotional/psychological aspects respectively. The total score is the sum of all item responses for total and dimension scores.
Time Frame: 12 weeks from baseline
Population: Mean of total score in the Minnesota Living with Heart Failure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Arm - Metoprolol Succinate.
Number analyzed (Participants) | 10
score on a scale
  Minnesota Living with Heart Failure scale at baseline | 74 (16)
  Minnesota Living with Heart Failure scale post treatment | 52 (18)

ADVERSE EVENTS:
Time Frame: Patients were monitored for AEs/SAEs for the duration of treatment (up to 12 weeks)
Description: Self reported AEs/SAEs
Arm/Group | Study Arm - Metoprolol Succinate.
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm - Metoprolol Succinate. (N=10)
Symptomatic hypotension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT05096884/Prot_SAP_000.pdf